CLINICAL TRIAL: NCT02116686
Title: ECG Derived Respiration for Automated Screening of Sleep Disordered Breathing in Chronic Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: OBS2014
Record Dates: First submitted 2014-04-10; First posted 2014-04-17 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure; Sleep Apnea Syndromes; Polysomnography
Keywords: chronic heart failure; Polysomnography; Sleep Apnea Syndromes; Electrocardiogram
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure patients with sleep apnea syndrom: For heart failure patients, a standard nocturnal in-home ventilatory polygraphic recordings were performed using an Embla device (Embla®, Broomfield, USA) and scored according to the America Academy of Sleep Medicine (AASM) recommendations (RemLogic® software, Broomfield, USA).
  Interventions: Device: ventilatory polygraphic recordings

INTERVENTIONS:
Device: ventilatory polygraphic recordings — Standard nocturnal in-home ventilatory polygraphic recordings were performed using an Embla device (Embla®, Broomfield, USA) and scored according to the AASM recommendations (RemLogic® software, Broomfield, USA).
  Other Names: Embla device (Embla®, Broomfield, USA); RemLogic® software, Broomfield, USA

SUMMARY:
The prevalence of sleep disordered breathing (SDB) reaches more than 50% in chronic heart failure patients (CHF). The main consequence is an increase risk of fatal and non-fatal cardiovascular events. A treatment by continuous positive airway pressure (CPAP) or adaptative servo-ventilation (ASV) reduces this risk. Nevertheless, 75% of severe SDB cases remains undiagnosed and untreated especially due to cost and time delay for polysomnography examination which is the gold standard for SDB diagnosis. Indeed, alternative methods are developed. Some methods, based on nocturnal ECG analysis showed promising results but they are not validated and adapted for cardiac population. Thus, the goal of present study is to test the accuracy of ECG derived respiration signal to screen SDB in a CHF population.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure
* left ventricular ejection fraction < 45%
* New York Heart Association (NYHA) index ≥ 2
* Sleep apnea syndrom confirmed by polysomnography

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease with maximal Respiratory Volume < 50%
* Resting oxygen saturation < 90%
* Continuous Positive Airway Pressure (CPAP) or Adaptive Servo-Ventilation treatment
* Life expectancy < 1 year for other medical reasons than heart failure
* Cardiac surgery
* Percutaneous transluminal coronary angioplasty
* Unstable angora during the 6 last months
* Implantation of a pacemaker or a defibrillator during the 6 last months
* Cerebrovascular accident or Transient Ischemic Attack during the 3 last months
* Restless legs syndrome
* Acute myocarditis or pericarditis during the 6 last months
* Valvular disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with sleep apnea syndrom
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | At patient polygraphic recording
  Standard nocturnal in-home ventilatory polygraphic recordings. The AHI is calculated only on nocturnal ECG analysis

SECONDARY OUTCOMES:
AHI in subgroup patient with sinusal rhythm | At patient polygraphic recording
AHI in subgroup with implanted pacemaker | At patient polygraphic recording
AHI in subgroup with atrial fibrillation | At patient polygraphic recording
AHI in subgroup with bundle branch block | At patient polygraphic recording

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ROCHE, MD PhD, Study Director — CHU de Saint-Etienne
Locations (2):
- France (2):
  - CHU de Grenoble, Grenoble
  - CHU de Saint-Etienne, Saint-Etienne